CLINICAL TRIAL: NCT03647423
Title: QUILT-3.091 NANT Chordoma Vaccine: A Randomized Phase 1b/2 Trial of the NANT Chordoma Vaccine vs. Radiation in Subjects With Unresectable Chordoma.
Brief Title: QUILT-3.091 NANT Chordoma Vaccine vs Radiation in Subjects With Unresectable Chordoma.
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial not initiated
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.091
Record Dates: First submitted 2018-08-09; First posted 2018-08-27 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2018-08

CONDITIONS: Chordoma; Unresectable Malignant Neoplasm
MeSH Terms: conditions — Chordoma | interventions — ALT-803; avelumab; Cetuximab; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Chordoma Vaccine: A randomized phase 1b/2 trial of the NANT chordoma vaccine vs. radiation in subjects with unresectable chordoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NANT Chordoma Vaccine (Experimental): A combination of agents will be administered to subjects in this study: Aldoxorubicin Hydrochloride HCI, ALT-803, ETBX-051, ETBX-061, GI-6301, haNK, avelumab, cetuximab, cyclophosphamide, SBRT.
  Interventions: Biological: Aldoxorubicin Hydrochloride; Biological: ALT-803; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-6301; Biological: haNK; Drug: Avelumab; Drug: Cetuximab; Drug: Cyclophosphamide
- Controlled Arm - Radiation (Active Comparator): SBRT
  Interventions: Radiation: SBRT

INTERVENTIONS:
Biological: Aldoxorubicin Hydrochloride — Aldoxorubicin Hydrochloride HCI
  Arms: NANT Chordoma Vaccine
Biological: ALT-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
  Arms: NANT Chordoma Vaccine
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury
  Arms: NANT Chordoma Vaccine
Biological: ETBX-061 — Ad5 [E1-, E2b-]-mucin 1 [MUC1]
  Arms: NANT Chordoma Vaccine
Biological: GI-6301 — Brachyury yeast
  Arms: NANT Chordoma Vaccine
Biological: haNK — haNK™, NK-92 [CD16.158V, ER IL-2]
  Arms: NANT Chordoma Vaccine
Drug: Avelumab — injection
  Other Names: BAVENCIO®
  Arms: NANT Chordoma Vaccine
Drug: Cetuximab — Injection
  Other Names: ERBITUX®
  Arms: NANT Chordoma Vaccine
Drug: Cyclophosphamide — Capsules
  Other Names: Cytoxan
  Arms: NANT Chordoma Vaccine
Radiation: SBRT — Stereotactic body radiation therapy
  Arms: Controlled Arm - Radiation

SUMMARY:
QUILT 3.091 Chordoma Vaccine: Phase 1B/2 NANT Chordoma Vaccine vs Radiation in Subjects with Unresectable Chordoma.

DETAILED DESCRIPTION:
The NANT Chordoma Vaccine regimen will be administered in 2 phases, an induction and a maintenance phase.

Subjects will continue induction treatment for up to 1 year. Those who have a confirmed complete response (CR) in the induction phase will enter the maintenance phase of the study. Subjects who experience ongoing stable disease (SD) or an ongoing partial response (PR) at 1 year may enter the maintenance phase at the Investigator's and Sponsor's discretion. Subjects may remain in the maintenance phase of the study for up to 1 year.

In the randomized component of the phase 2 portion of the study, the control arm will be treated with radiation according to established SoC protocols as determined by the Investigator.

In the phase 2 single-arm component of the study, subjects will be enrolled in the first stage of Simon's two-stage optimal design. If the study proceeds to the second stage of Simon's two-stage optimal design, additional subjects will be enrolled in the second stage.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
3. Histologically-confirmed recurrent or unresectable chordoma that would require radiation as a primary means for treatment.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Have at least 1 measurable lesion of ≥ 1.0 cm.
6. Must have a recent formalin-fixed, paraffin-embedded (FFPE) tumor biopsy specimen following the conclusion of the most recent anticancer treatment and be willing to release the specimen for prospective and exploratory tumor molecular profiling. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
7. Must be willing to provide blood samples prior to the start of treatment on this study for tumor molecular profiling and exploratory analyses.
8. Must be willing to provide a tumor biopsy specimen 8 weeks after the start of treatment for exploratory analyses, if considered safe by the Investigator.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non- sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Randomized component only - 11. Must be able to be classified into at least 1 of the below 3 categories: i. Recurred within 6 months after treatment, ii. Have metastatic disease, iii. Meet ≥ 4 of the histopathologic and immunohistochemical criteria: • Poorly differentiated histopathologic sub type, • Mitotic figures ≥ 3, • Apoptosis present. • Prominent nucleoli present, • Necrosis present, • Ki67 ≥ 6%, • p53 ≥ 25%

Single-arm component only 12. Must have progressed on or after radiation monotherapy in the randomized portion of the study OR been ineligible for the randomized portion but had progressed or experienced unacceptable toxicity on SoC prior to enrollment on the study.

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis,Addison's disease, or autoimmune disease associated with lymphoma).
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results: a. Absolute neutrophil count < 1,000 cells/mm^3, b. Uncorrectable grade 3 anemia (hemoglobin < 8 g/dL), c. Platelet count < 75,000 cells/mm^3, d. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome), e. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases), f. Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases), g. Serum creatinine > 2.0 mg/dL or 177 μmol/L, h. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication. Subjects with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
7. Serious myocardial dysfunction defined by ECHO as absolute left ventricular ejection fraction (LVEF) 10% below the institution's lower limit of predicted normal.
8. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
9. Positive results of screening test for human immunodeficiency virus (HIV).
10. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
11. Known hypersensitivity to any component of the study medication(s).
12. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
13. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
14. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
15. Participation in an investigational drug study or history of receiving any investigational treatment within 30 days prior to screening for this study, except for testosterone- lowering therapy in men with prostate cancer.
16. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
17. Concurrent participation in any interventional clinical trial.
18. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-31 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs), graded using the NCI CTCAE Version 4.03. | 9 weeks
  Phase 1b primary endpoint
Progression-free survival (PFS) by RECIST v1.1 | 1 years
  Phase 2 primary endpoint

SECONDARY OUTCOMES:
Objective response rate by RECIST v1.1 | 9 weeks
  Phase 1b secondary endpoint
Objective response rate by irRC | 9 weeks
  Phase 1b secondary endpoint
Progression-free survival (PFS) by RECIST v1.1 | 9 weeks
  Phase 1b secondary endpoint
Progression-free survival (PFS) by irRC | 9 weeks
  Phase 1b secondary endpoint
Overall survival | 9 weeks
  Phase 1b secondary endpoint
Disease control rate by RECIST v1.1 and irRC. | 1 year
  Phase 1b secondary endpoint
Disease control rate (confirmed complete response, partial response, or stable disease lasting for at least 2 months) by RECIST v1.1 and irRC. | 1 year
  Phase 1b secondary endpoint
Patient-reported outcomes of Chordoma cancer symptoms | 1 year
  Phase 1b secondary endpoint (by RECIST v1.1 and irRC and FACT-Hep questionnaire)
Progression-free survival (PFS) by irRC | 1 year
  Phase 2 secondary endpoint
Objective response rate by RECIST 1.1 | 1 year
  Phase 2 secondary endpoint
Objective response rate by irRC | 1 year
  Phase 2 secondary endpoint
Overall survival | 1 year
  Phase 2 secondary endpoint
Duration of response by RECIST and irRC | 1 year
  Phase 2 secondary endpoint
Disease control rate (confirmed complete response, partial response, or stable disease lasting for at least 2 months) by RECIST and irRC. | 1 year
  Phase 2 secondary endpoint
Patient-reported outcomes of Chordoma cancer | 1 year
  Phase 2 secondary endpoint
Incidence of treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs), graded using the NCI CTCAE Version 4.03. | 1 year
  Phase 2 secondary endpoint by (RECIST v1.1 and irRC and FACT-Hep questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: No